CLINICAL TRIAL: NCT04621344
Title: 30-DAY MORBIDITY, MORTALITY AND UNPLANNED HOSPITAL ADMISSIONS AFTER GUIDED-BRONCHOSCOPY AND ENDOSONOGRAPHY
Brief Title: Complications After Endosonography and Guided Bronchoscopy
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ST1
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Complication of Bronchoscopy
Keywords: Endosonography; Guided bronchoscopy; Complications; Hospital admission; Lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Guided bronchoscopy and/or endosonography — Endoscopic procedures aimed at sampling of intrathoracic lymph nodes or pulmonary lesions

SUMMARY:
The present study aims to investigate prospectively and systematically the direct and indirect complications occurring within 30 days after guided-bronchoscopy and/or endosonography. The results of the study should reliably help clarify further incidence, pattern, risk factors, and outcomes for both immediate and late complications associated with these key diagnostic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years,
* Indication to undergo bronchoscopy, endosonography, or both.
* Signed informed consent

Exclusion Criteria:

* Absolute contraindications to the bronchoscopic examination based on international guidelines [31].
* Platelet count <50000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication to guided bronchoscopy, endosonography, or both-
Sampling Method: Probability Sample
Enrollment: 701 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Incidence of severe complications | 30 days

SECONDARY OUTCOMES:
Overall incidence of complications | 30 days
Risk factors associated with severe complications | 30 days
Rate of unplanned hospital admissions | 30 days
Mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Trisolini, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli IRCS, Università Cattolica del Sacro Cuore
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No